CLINICAL TRIAL: NCT00173641
Title: The Role of Regulatory T Cell in Patients With Type 1 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700823
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-11-24 (Estimated); Status verified 2005-09

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: blood drawing

SUMMARY:
Evaluate the regulatory T cell function in patients with type 1 diabetes mellitus, and find the pathogenesis of this autoimmune disease.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1D) is an autoimmune disease characterized with T cell mediated destruction of pancreatic βcell. Dysregulated B and T cells were reported in the animal model. The loss of maintenance of immune homeostasis is thought to be major mechanism and result in persistence of autoreactive T cell in the periphery. Therapies which modulate the immune dysfunction may be helpful for the patients of T1D.

Immune homeostasis means a balance between the responses that control infection and tumor growth and reciprocal responses that prevent inflammation and autoimmune disease. CD4+ CD25+ regulatory T cells (Tregs) are critical to maintain such functions. Their actions can be through cell-to-cell contact or bystander effect. The specific markers of Tregs include CD25 molecule (IL-2 receptorαchain), Foxp3 (forkhead-winged helix transcription factor). The Foxp3 is a transcription factor that controls some genes encoding Tregs associated molecules, such as CD25, CTLA-4 and GITR.

The previous studies of modulation of Tregs in T1D show positive results in animal model. But the relative sizes of CD4+CD25+ population in human are still controversial. Our hypothesis is that the imbalance of Tregs and autoreactive T cells is the pathogenesis of T1D. Therefore, we used flow cytometry to determine the number of CD4+CD25+ Tregs population and quantitative real-time PCR to assay the expression of Foxp3, CLTA-4, GITR in patients with different stages and normal control. Besides, autoantibodies to GAD65 is associated with T1D in 60-80% patients. It is a marker of autoimmune diabetes. We anticipated that the realization of Tregs functions in patients of T1D will help our further guide of immunotherapy of patients with T1D and other autoimmune disease.

ELIGIBILITY:
Inclusion Criteria:

* pediatric type 1 DM

Exclusion Criteria:

-

Ages: 1 Month to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150
Dates: Start 2005-09; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ching Tung, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Putnam AL, Vendrame F, Dotta F, Gottlieb PA. CD4+CD25high regulatory T cells in human autoimmune diabetes. J Autoimmun. 2005 Feb;24(1):55-62. doi: 10.1016/j.jaut.2004.11.004. Epub 2005 Jan 12. PMID 15725577